CLINICAL TRIAL: NCT05155293
Title: A Randomized, Double-masked, Parallel-group, Multicenter Clinical Study to Evaluate the Efficacy and Safety of AVT06 Compared With EU-Eylea® in Subjects With Neovascular (Wet) Age-related Macular Degeneration (ALVOEYE)
Brief Title: Clinical Study to Compare Efficacy and Safety of AVT06 and EU-Eylea (ALVOEYE)
Acronym: ALVOEYE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT06-GL-C01
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Neovascular (Wet) AMD
Keywords: Macular Degeneration; Retinal Degeneration; Aflibercept
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT06 (proposed aflibercept biosimilar) (Experimental): Patients will receive 1 IVT injection of AVT06 every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  Interventions: Drug: AVT06 (proposed aflibercept biosimilar)
- Eylea® (Aflibercept) (Experimental): Patients will receive 1 IVT injection of Eylea® every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  Interventions: Drug: Eylea® (Aflibercept)

INTERVENTIONS:
Drug: AVT06 (proposed aflibercept biosimilar) — Patients will receive IVT injections of AVT06
  Arms: AVT06 (proposed aflibercept biosimilar)
Drug: Eylea® (Aflibercept) — Patients will receive IVT injections of Eylea®
  Arms: Eylea® (Aflibercept)

SUMMARY:
This is a randomized, double-masked, parallel-group, multicenter, therapeutic equivalence study evaluating the efficacy, safety, and immunogenicity of AVT06 compared with Eylea in subjects with neovascular (wet) AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥50 years of age, at the time of signing the informed consent.
* Subjects must be diagnosed with neovascular (wet) AMD in the study eye.
* Subjects must have active, treatment naïve, subfoveal CNV lesions secondary to neovascular (wet) AMD.
* Willingness and ability to undertake all scheduled visits and assessments.

Exclusion Criteria:

* Any prior systemic treatment with anti-VEGF therapy
* Any condition that, in the Investigator ́s opinion, can interfere with full participation in the study, including administration of the study treatment and attending required visits; can pose a significant risk to the participant, or interfere with interpretation of study data
* Prior treatment with any investigational drugs within 30 days or 5 half-lives (whichever is longer) of the previous investigational treatment before initiation of the study treatment or concomitant enrollment in any other clinical study involving an investigational study treatment
* Subjects not suitable for participation, whatever the reason, as judged by the Investigator, including medical or psychiatric conditions, or participants potentially at risk of noncompliance to study procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 8 in Best-corrected Visual Acuity (BCVA) | Week 8

CONTACTS AND LOCATIONS:
Locations (6):
- Nemocnicni lekarna Sokolov, Sokolov, Czechia
- JSC Evex Medical Corporation, Tbilisi, Georgia
- Keneikai Hayashi Eye Hospital, Fukuoka, Japan
- Latvia (2):
  - Riga East University Hospital Clinical Centre "Bikernieki", Riga
  - Pauls Stradins Clinical University Hospital SLLC, Riga
- Fakultna Nemocnica Trencin, Trenčín, Slovakia

REFERENCES:
- [Derived] Agostini H, Baumane K, Balciuniene VJ, Ozols K, Soni R, Hamdi S, Cirillo S, Rai M, Otto H, Leutz S, Sattar A, Berti F. A randomized, double-masked parallel-group, multicenter clinical study evaluating the efficacy and safety of the biosimilar candidate AVT06 compared to the reference product aflibercept in participants with neovascular age-related macular degeneration. Expert Opin Biol Ther. 2025 Jul;25(7):773-787. doi: 10.1080/14712598.2025.2519531. Epub 2025 Jun 17. PMID 40512025